CLINICAL TRIAL: NCT04411745
Title: Capturing Early Events in Human Parturition Based on Whole-transcriptome Analysis of Maternal Blood Before and After Spontaneous Onset of Labor at Term
Brief Title: Capturing Early Events in Human Parturition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tak Yeung LEUNG, Professor, Chinese University of Hong Kong
Other Study IDs: 2015.659
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Parturition; Precipitate
Keywords: transcriptome
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturition: Healthy women who are carrying a healthy singleton pregnancy, but have not yet gone to labor at 40 weeks of gestation or who are at term and admitted to hospital for any sign of labor.
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study

SUMMARY:
This is a prospective observational study on normal singleton pregnant women who have no sign of labor at 40 weeks of gestation or pregnant women who admitted to hospital for any sign of labor at term, aiming to identify labor-associated markers.

DETAILED DESCRIPTION:
The mechanisms that instigate human parturition have not been completely understood, though hypotheses such as 'functional progesterone withdrawal' and inflammatory signaling have been proposed. Researchers including our group have previously identified panels of genes which were differentially expressed between placentas obtained after spontaneous birth and those after elective cesarean delivery. However, such findings obtained after birth could only reflects the late changes in parturition. Similar findings in other gestational tissues, such as fetal membranes, amniotic fluids, myometrial biopsies are available, but these sample types cannot be readily collected until delivery.

Thus, we propose to explore biomarkers in maternal blood with a view to developing any useful analytes for predicting labor.

ELIGIBILITY:
Inclusion Criteria:

Healthy women who are carrying a healthy singleton pregnancy, but have not yet gone to labor at 40 weeks of gestation or who are at term and admitted to hospital for any sign of labor are invited to join the study.

Exclusion Criteria:

* Any obstetric contraindications for undergoing labor or vaginal delivery (e.g. placenta previa, cephalo-pelvic disproportion, macrosomia, previous classical cesarean section or uterine tear, etc).
* Any maternal or fetal complications that require immediate or early delivery (e.g. pre-eclampsia, abruption placenta, fetal distress, rupture of membranes, in utero death, etc).
* Any maternal or fetal complications that make vaginal birth an unfavorable choice (e.g. fetal growth restriction, fetal compromise or distress, etc).
* Any conditions that are known to affect the onset of labor (e.g. anencephaly).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Healthy women who are carrying a healthy singleton pregnancy, but have not yet gone to labor at 40 weeks of gestation or who are at term and admitted to hospital for any sign of labor.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
RNA gene expression | Between 36 and 41 weeks of gestation
  Peripheral blood samples will be taken for RNA gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Tak Yeung LEUNG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong